CLINICAL TRIAL: NCT03642886
Title: The Use of Prescribed Detraining to Decrease Atrial Fibrillation Burden and Symptoms in Athletes.
Brief Title: Detraining on Atrial Fibrillation
Acronym: DAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiology Research UBC (Other)
Responsible Party: Principal Investigator, James McKinney, Research Director at SportsCardiologyBC, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: InterventionalCR
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: In adjudication of arrhythmia events the adjudicators would not know if the participants have been randomized to the detraining or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continued Strenuous Exercise (No Intervention): Continued strenuous athletics (no reduction in training volume) - athletes will be asked to document their activity and be fitted with an activity monitor during the run-in period and intervention period
- Prescribed Detraining (Experimental): Detraining period of 8-weeks which is defined as:
  1. a 75% decrease in the amount of exercise (from baseline)
  2. a 50% decrease in the intensity of exercise as measured in METS (from baseline)
  3. Mitchell Classification classes 1A, 2A, 2B of activity are permitted
  Interventions: Behavioral: Prescribed Detraining

INTERVENTIONS:
Behavioral: Prescribed Detraining — Detraining is the deliberate act of reducing volume of exercise to observe subsequent changes in cardiac indices over time or the partial or complete loss of training of induced anatomical, physiological and performance adaptions. Detraining is primarily employed as a diagnostic tool to help differentiate Athletes' heart from cardiac pathology.
  Arms: Prescribed Detraining

SUMMARY:
This study will examine the effect of detraining as a clinical tool to prevent recurrence of lone paroxysmal atrial fibrillation (AF) and improve quality of life. Persons who engage in endurance activity with AF will be randomly assigned to undergo an 8-week period of detraining or encouraged to maintain their current level of exercise. Participants will receive a handheld device called AliveCor that can record an electrical tracing of the heart rhythm by pressing down with ones' thumbs. The amount of arrhythmia and symptoms will be recorded. The research team hypothesizes that among athletes with lone AF, an 8-week period of detraining will not affect atrial fibrillation recurrence or quality of life.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common tachyarrhythmia amongst athletes. Atrial fibrillation is associated with poor subjective health among Masters athletes, and negatively interferes with athlete's sporting activities. The decrease in physical performance during AF episodes is attributed to the loss of atrial contribution to cardiac output related to irregular and decreased diastolic filling, and loss of sympathetic and parasympathetic control over heart rate.

There is a paucity of studies that examine the role of exercise in the treatment of atrial fibrillation among athletes. Detraining is the deliberate act of reducing volume of exercise to observe subsequent changes in cardiac indices over time or the partial or complete loss of training of induced anatomical, physiological and performance adaptions. Detraining is primarily employed as a diagnostic tool to help differentiate Athletes' heart from cardiac pathology. The role of detraining as a therapeutic modality is ill-defined and not well studied. There is a dearth of studies that examine the role of exercise in the treatment of atrial fibrillation among athletes. To date, only two observational studies (Furlanello and Hoogsteen) have suggested detraining as a potential treatment for AF among athletes. It is important to note the limitations of these studies: 1) observational study design 2) athletes were not systematically instructed to decrease exercise volume or 'detrain' 3) AF was not objectively assessed 4) pre and post measures of QOL were not recorded AF. Hoogsteen et al., surveyed 30 athletes about exercise and AF symptomatology at the time of diagnosis and 9 years later. At the time of the survey 30% of athletes noted a reduction in bouts of AF with a decrease in sporting activity. However, 43% of the athletes did not notice any relationship between reduction in activity and AF recurrence. This study was limited by the small sample size, selection bias due to symptomatic athletes responding, and AF recurrence based solely on subjective responses.

Detraining has been shown to decrease premature ventricular contractions (PVCs) and non-sustained ventricular tachycardia (NSVT) burden amongst elite athletes. After a 3-month detraining period, PVCs and NSVT decreased by eighty and ninety percent, respectively. The same group of athletes experienced a prolonged suppression of PVCs and NSVT at 1-year after retraining. While detraining is often suggested to athletes with AF, there is little evidence to support this practice. To date, only small case series and individual case reports exist.

This study aims to examine the effect of detraining as a clinical tool to prevent recurrence of lone paroxysmal AF (with no traditional AF risk factors and a structurally normal heart) and improve quality of life. Persons who engage in endurance activity with AF will be randomly assigned to undergo a 10-week period of detraining or encouraged to maintain their current level of exercise. Participants will receive a (1x 2.5 inch) handheld device called AliveCor that can record an electrical tracing of the heart rhythm by pressing down with ones' thumbs. The amount of arrhythmia and symptoms will be recorded. The research team hypothesizes that among athletes with lone AF, a 10-week period of detraining will not affect atrial fibrillation recurrence or quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60
2. Paroxysmal AF (eligible subjects must have had >1episode of AF within the last 12 months)
3. Performs prolonged regular sessions of strenuous practice (≥6h/week with intensity greater than 60% of maximum heart rate for at least 6 months prior)
4. Preserved ejection fraction (≥ 55%) with an absence of structural heart disease (hypertrophic cardiomyopathy, valvular heart disease, hypertensive heart disease)

Exclusion Criteria:

1. BMI > 25 kg/m2
2. Hypertension as per 2016 Canadian Hypertension Education Program Guidelines[52]
3. Diabetes
4. Structural heart disease
5. Obstructive sleep apnea
6. Metabolic abnormalities (hyperthyroidism, pheochromocytoma)
7. Pericarditis
8. Coronary artery disease (defined as history of myocardial infarction, angina, q-waves on resting ECG, perfusion defect on nuclear scan, wall-motion abnormality on echocardiogram).
9. Pre-excitation, Brugada syndrome, Long QT syndrome, arrhythmogenic cardiomyopathy or catecholaminergic polymorphic ventricular tachycardia
10. Use of performance-enhancing agents
11. Implanted cardiac pacemaker or defibrillator
12. A concurrent period of involuntary deconditioning

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of atrial fibrillation (AF) episodes | 0-32 weeks
  Determine the effectiveness of systematic detraining on AF episodes (the number of AF AliveCor transmissions over the total number of daily transmissions (ECGaf/ECGtotal))
Symptomatic palpitations | 0-32 weeks
  The number of patient reported symptomatic palpitations that correspond with documented atrial fibrillation (some participants may be experiencing AF but may not actually be symptomatic)

SECONDARY OUTCOMES:
AF symptom severity | Taken at 0, 8, and 32 weeks
  AF symptom severity score at baseline, after completion of 8 weeks of either control or detraining, and at completion of 24 weeks of post-intervention monitoring. Measured using the Cardiovascular Society Severity of Atrial Fibrillation (SAF) Scale which identifies the presence of symptoms, the association of symptoms with AF, and the affect these symptoms have on the patients functionality. Based on the patient's responses, an SAF class of 0-4 is assigned. Class 0 refers to a patient who is asymptomatic with respect to AF while a class 4 patient has symptoms attributed to AF that have a severe effect on the patient's general quality of life.
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) score | Taken at 0, 8, and 32 weeks
  AFEQT score at baseline, after completion 8 weeks of either control detraining, and at completion of 24 weeks of post-intervention monitoring. The questionnaire is comprised of 12 questions (4 focused on the extent to which patients are bothered by symptoms associated with AF, 2 focused on the extent to which patients feel limited in their daily life due to AF, and 6 focused on the difficulty that patients feel in doing daily activities due to AF) responded to on a 7-point scale where 1 represents being not at all bothered, limited or experiencing no difficulty, and 7 represents being extremely bothered, limited or experiencing extreme difficulty.
General quality of life | Taken at 0, 8, and 32 weeks
  General QOL will be assessed using the 12-item Short Form Health Survey (SF-12) at baseline, after completion of 8 weeks of either control or detraining, and at completion 24 weeks of post-intervention monitoring. The SF-12 is a validated survey that was designed as a condensed version of the RAND 36-item Short Form Health Survey Instrument (SF-36) and provides two scores: physical and mental health composite scores (PCS & MCS). The scores are computed on a scale from 0 to 100 where a score of zero represents the lowest level of health measured and 100 represents the highest level of health. For both the PCS and MCS, the responses from the 12 questions are combined and scored in such a way that they compare to an American national norm of 50.0 (with a standard deviation of 10.0).
Hospitalizations/emergency room visits | 0-32 weeks
  Number of hospitalizations/emergency room visits over the course of the study will be recorded.
DC cardioversions | 0-32 weeks
  The number of DC cardioversions received by the participants throughout the course of the study will be recorded.
Percent referred for AF ablation | 0-32 weeks
  The percent of participants referred for AF ablation throughout the course of the study will be recorded. (number of participants referred for AF ablation/total number of participants)
Initiation of anti-arrhythmic drug therapy | 0-32 weeks
  The number of participants who initiate anti-arrhythmic drug therapy throughout the course of the study will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: James McKinney, MD, Principal Investigator — University of British Columbia Department of Medicine
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada